CLINICAL TRIAL: NCT05574387
Title: Metformin, The Biguanide Derivative, as Adjuvant Therapy in Patients With Ulcerative Colitis Treated With Mesalamine
Brief Title: Metformin as Added on Therapy in Patients With Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Principal Investigator Mostafa Mahmoud Bahaa El-Dien Pharmacy Practice Department- Horus University (Unknown)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6/2022
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will take mesalamine 1 g three times daily
- Metformin group (Active Comparator): This group will take mesalamine 1 g three times daily plus metformin 500 mg two times daily
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is an antidiabetic biguanide drug that acts by promoting glucose uptake and utilization in the liver.Recent studies proved that metformin could reduce colonic inflammation by AMPK-mediated inhibition of p38 mitogen-activated protein kinase (MAPK)
  Arms: Metformin group

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease that is marked by increased intestinal motility and bloody diarrhea. The clinical value of existing therapeutic strategies of UC, including glucocorticoids, anti-tumor necrosis factor α (TNF-α), mesalamine, and thiopurines is still limited. Therefore, the discovery of new therapeutic approaches is essential to improve the effectiveness of the treatment.Adenosine monophosphate (AMP)-activated protein kinase (AMPK) is a conserved fuel-sensing enzyme that plays an important role in the regulation of cellular metabolism where it increases glucose and fatty acids uptake and activates the oxidation process to improve the cellular energy utilization

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years Both males and females will be included Negative pregnancy test and effective contraception Mild and moderate UC patients diagnosed and confirmed by the endoscope

Exclusion Criteria:

- Breastfeeding Significant liver and kidney function abnormalities Diabetic patients Colorectal cancer patients Patients with severe UC Patients taking rectal or systemic steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in HRQL through changes in inflammatory bowel disease questionnaire (IBDQ) score and change in mayo scores | 6 months
  The IBDQ includes 32 questions, The questions are grouped into four categories: bowel symptoms (B), systemic symptoms (S), emotional function (E), and social function (SF). Response options are consistently presented as seven-point scales, scores range from 32-224.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt